CLINICAL TRIAL: NCT05022238
Title: Hotspots, Households and Hospitals: Enhanced Drug-resistant Tuberculosis Case Finding in Namibia
Acronym: H3TB
Status: Recruiting | Type: Observational
Sponsor: University of Namibia (Other)
Collaborators: UK Medical Research Council (MRC) (Unknown); European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government); Research Center Borstel (Other); Imperial College London (Other); University of Stellenbosch (Other); National Taiwan University (Other); Namibian National Tuberculosis and Leprosy Programme (NTLP) (Unknown); UK Foreign, Commonwealth & Development Office (FCDO) (Unknown)
Responsible Party: Principal Investigator, Mareli Claassens, Associate research professor, University of Namibia
Other Study IDs: HGC/611/2021
Record Dates: First submitted 2021-08-10; First posted 2021-08-26 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-05

CONDITIONS: Tuberculosis, Multidrug-Resistant
Keywords: case-finding; Namibia
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Sputum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Poor case management, pharmacokinetic variability and on-going transmission have fostered the drug-resistant tuberculosis (DR-TB) epidemic leading to a global estimated number of >500,000 new multidrug resistant (MDR) TB cases per year, of which roughly 10% are extensively drug resistant (XDR). Namibia is a high TB burden country with an incidence rate of 446/100,000 in 2016; about 11,000 new cases per year. 3.9% of new cases and 8.7% of previously treated cases have MDR-TB. Whole genome sequencing (WGS) has recently been applied to interrogate the complete genetic code of Mycobacterium tuberculosis (Mtb) strains. WGS can be used to infer relationships between identified strains as well as determine genomic variations involved in resistance development.

The specific aims of the H3TB study are to: (i) characterise the DR-TB epidemic, in terms of clinical, epidemiological, geospatial, social network and laboratory data, to identify transmission hotspots in three regions of Namibia, (ii) evaluate the feasibility of targeted case finding intervention strategies to improve DR-TB control in highly affected populations and (iii) develop a transmission model to investigate the potential impact of the case finding intervention strategies on DR-TB incidence in Namibia.

A prospective surveillance study started in January 2020, which includes all DR-TB cases in Namibia, and which will nest H3TB. Data collection tools and other study implementation tools have been designed and implemented. The study team is working in close collaboration with the National Institute of Pathology, where all DR-TB cases from the country are registered, to ensure all possible cases are captured. This is important for the identification of transmission hotspots.

After HREC and MOHSS approval, individuals with GeneXpert® MTB/RIF rifampicin-resistant samples and a positive Mtb culture from three regions in Namibia will be included in a transmission hotspot identification study. Preliminary data have shown that DR-TB clusters exist in these regions. Clinical, epidemiological, geospatial, social network and laboratory data (GeneXpert® MTB/RIF, culture, drug sensitivity tests) will be collected. WGS capacity has been established at the UNAM research laboratory, where WGS will be performed on the samples of H3TB participants; results will be validated at the Research Center Borstel in Germany. These study results in conjunction with a systematic review and meta-analysis will inform the design of case finding interventions which will be evaluated through a mixed-methods feasibility study conducted at high transmission areas (hotspots, households and hospitals). Data from these studies and the TB programme will be used to develop the model which will include a health economics component.

The study will strengthen DR-TB diagnosis, surveillance and control, inform DR-TB case finding policy in Namibia and regionally, inform resource allocation by identifying high transmission areas and create preliminary data to design a large scale DR-TB case finding intervention.

ELIGIBILITY:
Inclusion Criteria:

* All cases diagnosed with drug-resistant TB in Namibia, in three regions of Khomas, Otjozondjupa and Ohangwena will be included for the first outcome. For the second outcome, all household members of DR-TB cases will be included; all hospital visitors to DR-TB cases will be included and community members at transmission hotspots will be included.

Exclusion Criteria:

* Anyone who does not give consent to participate.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: For the first outcome, the study population is all DR-TB cases in three regions of Namibia, diagnosed by the National Institute of Pathology (GeneXpert Ultra Rifampicin resistant) over 18 months.
  For the second outcome, all household contacts of DR-TB cases in the three regions is the study population, as well as DR-TB patients' hospital visitors and community members at transmission hotspots.
Sampling Method: Non-Probability Sample
Enrollment: 2100 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Identification of drug-resistant tuberculosis transmission hotspots in Namibia | 18 months
  Finding DR-TB transmission hotspots through whole genome sequencing (WGS), social network and shared space analyses, and geospatial analyses. WGS, social network and shared space data, and geospatial data, will be triangulated to identify transmission hotspots.
Feasibility study of three interventions to enhance drug-resistant TB case finding in Namibia, measured with a questionnaire | 24 months
  Evaluating the acceptability, yield and cost of three interventions, viz., finding cases in community transmission hotspots, in drug-resistant tuberculosis hospitals, and in households of drug-resistant tuberculosis patients, in three regions of Namibia
Transmission model | 12 months
  Using programmatic and data from outcomes 1 and 2 to develop and calibrate transmission model to look at the impact of scale-up of interventions

CONTACTS AND LOCATIONS:
Overall Officials: Mareli Claassens, PhD, Principal Investigator — University of Namibia
Locations (1):
- University of Namibia, Windhoek, Namibia

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared after the acceptance for publication of the main findings from the final dataset by researchers' efforts if a data transfer agreement is made between the custodians of the data (the H3TB study team) and other researchers, that: (i) data will be used only for research purposes, (ii) proper technological measures will be used to ensure data security, (iii) no effort will be made to identify study participants, (iv) data will be destroyed after the agreed analyses and (v) the data source will be acknowledged.
  The sequencing data will be made available on ReSeqTB or a similar platform. The other data will be stored locally at UNAM in a tailored database and made available by researchers' efforts. These data include individual-level information on health status (e.g., TB and HIV infection status) which cannot be made publicly available.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Once the primary analyses are complete, manuscripts submitted and final reports submitted to funding agencies.